CLINICAL TRIAL: NCT05028452
Title: Carer eSupport: Rationale and Design of an Internet-based Support for Informal Caregivers of Individuals With Head and Neck Cancer
Brief Title: Feasibility of Internet Based Support (Carer eSupport) for Informal Caregivers of Patients With Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Cancer Society (Other); Uppsala University Hospital (Other); Region Västerbotten (Other Government); Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Carer eSupport
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Caregivers; Head and Neck Cancer; Feasibility Study
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Single group posttest only design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet based support (Other): Internet based support for informal caregivers to individuals who are undergoing treatment for head and neck cancer.
  Interventions: Other: Internet based support

INTERVENTIONS:
Other: Internet based support — Carer eSupport is designed to prepare informal caregivers for caregiving, to decrease caregiver burden and prevent a deteriorated health.
  Other Names: Carer eSupport

SUMMARY:
Informal caregivers to patients with head and neck cancer report that they are unprepared for caregiving, that they experience a high caregiver burden and a deteriorated health. The aim is to develop an internet based intervention for informal caregivers of individuals with head and neck cancer and evaluate the feasibility and acceptability of the intervention. The internet based intervention (Carer eSupport) will be based on scientific evidence, established theoretical frameworks and focus groups with caregivers and health care professionals. The feasibility and acceptability of Carer eSupport will be evaluated by 30 caregivers who will have access to Carer eSupport during one months. The feasibility and acceptability of Carer eSupport will be evaluated with quantitative and qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregivers (defined by the patients) to patients with head and neck cancer who are about to start treatment, undergoing treatment or have completed treatment within the past month.

Exclusion Criteria:

* Confusion or dementia, inability to understand, speak or read Swedish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Inclusion rate | 4 months
  The proportion of caregivers who give informed consent for participation
Utilization of Carer eSupport | 2 months
  The proportion of included caregivers who take use of Carer eSupport
Attrition | 3 months
  The proportion of included caregivers who withdraw from the study
Completion of questionnaires | 3 months
  The proportion of included caregivers who complete questionnaires
Perceived feasibility | Within 1 months after completion of testing Carer eSupport.
  Qualitative data from semi-structured individual interviews exploring perceived feasibility of Carer eSupport.
Perceived acceptability | Within 1 months after completion of testing Carer eSupport.
  Qualitative data from semi-structured individual interviews exploring perceived acceptability of Carer eSupport.

SECONDARY OUTCOMES:
The Preparedness for caregiving scale | Assessed at baseline and at 1 months after access to Carer eSupport
  A brief 8-item self-report measure assessing preparedness for caregiving, a potential primary outcome in a future randomized controlled trial.
Caregiver´s burden scale | Assessed at baseline and at 1 months after access to Carer eSupport.
  A 22-item self-report measure assessing caregiver burden, a potential primary outcome in a future randomized controlled trial.
Short Form Health Survey (SF-36), v2. | Assessed at baseline and at 1 months after access to Carer eSupport.
  A 36-item self-report measure assessing self-perceived health, a potential secondary outcome in a future randomized controlled trial.
The Depression Anxiety Stress Scale-21 | Assessed at baseline and at 1 months after access to Carer eSupport.
  A 21-item self-report measure assessing depression, anxiety, and stress, a potential secondary outcome in a future randomized controlled trial.
The Multidimensional fatigue inventory | Assessed at baseline and at 1 months after access to Carer eSupport.
  A 20-item self-report measure assessing five dimensions of fatigue, a potential secondary outcome in a future randomized controlled trial.

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta Johansson, Docent, Principal Investigator — Uppsala University, Department of Immunology, Genetics and pathology
Locations (4):
- Sweden (4):
  - Örebro University Hospital, Örebro, Blekinge Län
  - Uppsala university hospital, Uppsala, Uppsala County
  - Norrland University Hospital, Umeå, Västerbotten County
  - Sahlgrenska university hospital, Gothenburg, Västra Götaland County

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers, since this is a feasibility study.

REFERENCES:
- [Derived] Langegard U, Cajander A, Carlsson M, von Essen L, Ahmad A, Laurell G, Tiblom Ehrsson Y, Johansson B. Internet-based support for informal caregivers to individuals with head and neck cancer (Carer eSupport): a study protocol for the development and feasibility testing of a complex online intervention. BMJ Open. 2022 May 27;12(5):e057442. doi: 10.1136/bmjopen-2021-057442. PMID 35623759